CLINICAL TRIAL: NCT00533286
Title: Do Benzodiazepines Improve the Outcome of Mechanical Physiotherapy for Lumbar Disk Prolapse: a Prospective Randomized Clinical Trial
Brief Title: Do Benzodiazepines Improve the Outcome of Mechanical Physiotherapy for Lumbar Disk Prolapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKF 57-0-0
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-09

CONDITIONS: Pain; Disability; Paresis
Keywords: physiotherapy; Tuebingen concept; benzodiazepines; muscle relaxants; disc herniation
MeSH Terms: conditions — Pain; Paresis; Muscle Hypotonia; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): placebo (2 tablets daily)
  Interventions: Drug: benzodiacepine
- B (Experimental): diazepam (2 x 5 mg)
  Interventions: Drug: benzodiacepine

INTERVENTIONS:
Drug: benzodiacepine — diazepam (2 x 5 mg/ die)

SUMMARY:
Sixty patients were randomized to receive either placebo or diazepam in addition to mechanical physiotherapy and analgesics for the first 7 days of conservative treatment of clinically and radiologically confirmed lumbar disk prolapse

ELIGIBILITY:
Inclusion Criteria:

* sciatica without or with neurological deficit attributable to lumbar disc prolapse
* CT or MRI confirmation of lumbar disc prolapse
* informed consent

Exclusion Criteria:

* bladder or bowel disturbance
* acute (< 24 h) development of paresis grade 1 or plegia
* taken benzodiazepines for more than 2 weeks
* history of benzodiazepine intolerance
* prior surgery for disc prolapse, or prior trauma to the vertrebral column

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
(i) median extent of reduction of referred pain | 7 days

SECONDARY OUTCOMES:
median duration of inability to work after discharge | one year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Prof., Principal Investigator — Department of General Neurology, University of Tuebingen Medical School, Tuebingen, Germany